CLINICAL TRIAL: NCT06718192
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Bleomycin and Cryotherapy in Treating Plantar Warts.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-206
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Verruca Plantaris
Keywords: verruca plantaris; Bleomycin; cryotherapy; efficiency; security
MeSH Terms: interventions — Bleomycin; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bleomycin Group (Active Comparator)
  Interventions: Other: Bleomycin injection
- cryotherapy (Other)
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Bleomycin injection — Wart injection (0.2 mL <5 mm; 0.5 mL 5-10 mm; 1ml for >10 mm) were injected at a depth of 1.5mm, diluted with normal saline at a concentration of 3u/ml=3mg/ml, and the maximum amount of each wart was 1ml until the wart turned white
  Arms: Bleomycin Group
Other: Cryotherapy — The wart was frozen by liquid nitrogen until a circle of frozen tissue appeared around the wart for about 10s, with an interval of 30s, for a total of 2 times
  Arms: cryotherapy

SUMMARY:
To evaluate the efficacy of bleomycin and cryopreservation in the treatment of plantar verruca by dermoscopy and explore the influencing factors. Compare the safety, economic burden and impact on quality of life of the two treatments

DETAILED DESCRIPTION:
Our research aims to evaluate and compare the effectiveness of bleomycin and cryotherapy in treating plantar warts. First, we enrolled patients according to eligibility criteria. Second, the patients were assigned to two groups randomly. One is Bleomycin Group and the other is Cryotherapy Group which means two -group-patients were received different therapies. Thirdly, we compared the efficiency of two groups by using dermoscopy. Finnally, we used statistical analysis to analyze the research data and draw the experimental conclusions.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years old, gender is not limited; Consistent with the diagnosis of plantar warts; Volunteer for treatment and sign informed consent; Consent to photograph the lesion; The treatment target area can be selected (the target area must meet the following conditions: The distance between adjacent warts in the target area is >0.5cm; The diameter of a single wart in the target area is ≤1.5cm, and/or the diameter of a wart mass is ≤1.5cm; The number of total warts/wart masses in the target area is ≤10).

Exclusion Criteria:

Patients who can't sign informed consent; Had previously received local treatment for common warts within 1 month; hiv-positive patient; Pregnant and lactating women; Has peripheral vascular disease; Allergic to bleomycin; People who are severely immunocompromised, or who are taking immunosuppressive drugs; Mental illness or cognitive incapacity; Other conditions deemed unsuitable for inclusion, such as inability to cooperate with follow-up, were considered by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
the rate of warts complete clearance | 2 weeks after treatment endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No